CLINICAL TRIAL: NCT00232245
Title: Use of Fish Oils to Reduce the Frequency and Duration of Episodes of Atrial Fibrillation in Patients With Paroxysmal Atrial Fibrillation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.216
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil (Experimental): Patients prescribed 6g/day of fish oil containing total 1.8 g of EPA+DHA in a 1.5:1 ratio
  Interventions: Drug: Fish oil
- Control (No Intervention): No fish oil exposure

INTERVENTIONS:
Drug: Fish oil
  Arms: Fish oil

SUMMARY:
The purpose of this study is to investigate whether fish oil supplements may reduce the frequency and duration of paroxysmal atrial fibrillation episodes.

Atrial fibrillation is a heart condition which effects a large percentage of the population .

Atrial fibrillation is a condition frequently experienced by people who have had pacemakers inserted .

Certain Pacemakers have sophisticated monitoring features that are able to recognise episodes of atrial fibrillation.

Fish oil supplements may be of benefit to patients with heart problems.Recent evidence suggests that fish oils may be beneficial to patients with rhythm disturbances.

By interrogating pacemakers this study will investigate the effect of fish oil supplements on the frequency and duration of episodes of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had at least 2 previous episodes of atrial fibrillation and an implanted pacemaker.

Exclusion Criteria:

* Patients with chronic atrial fibrillation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Atrial tachycardia and atrial fibrillation burden | 18 months

SECONDARY OUTCOMES:
Frequency and duration of atrial tachycardia/fibrillation episodes | 18 months

OTHER OUTCOMES:
Safety and tolerability of fish oil | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sparks, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Kumar S, Sutherland F, Stevenson I, Lee JM, Garg ML, Sparks PB. Effects of long-term omega-3 polyunsaturated fatty acid supplementation on paroxysmal atrial tachyarrhythmia burden in patients with implanted pacemakers: results from a prospective randomised study. Int J Cardiol. 2013 Oct 9;168(4):3812-7. doi: 10.1016/j.ijcard.2013.06.030. Epub 2013 Jul 26. PMID 23890856